CLINICAL TRIAL: NCT01836835
Title: Case-cohort Validation Study of Pregnancy Unique Questionnaire of Emesis (PUQE) in Norwegian
Brief Title: Pregnancy Specific Nausea Questionnaire (PUQE) Translated and Tested in Norwegian
Acronym: PUQE-N
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/465
Record Dates: First submitted 2013-04-08; First posted 2013-04-22 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Hyperemesis Gravidarum
Keywords: Hyperemesis gravidarum; Pregnancy; Nausea; Nutritional status; Questionnaire; Case-control
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hyperemesis gravidarum: Women diagnosed with hyperemesis gravidarum admitted to hospital Pregnancy Unique Questionnaire of Emesis (PUQE) and 24 hours self-reported nutritional intake form administered
  Interventions: Other: Pregnancy Unique Questionnaire of Emesis (PUQE); Other: 24 hours self-reported nutritional intake form
- Healthy pregnant women: Women with presumed normal pregnancy Pregnancy Unique Questionnaire of Emesis (PUQE) and 24 hours self-reported nutritional intake form administered
  Interventions: Other: Pregnancy Unique Questionnaire of Emesis (PUQE); Other: 24 hours self-reported nutritional intake form

INTERVENTIONS:
Other: Pregnancy Unique Questionnaire of Emesis (PUQE) — For hyperemesis gravidarum patients the Pregnancy Unique Questionnaire of Emesis (PUQE) (3 questions regarding the amount of nausea and vomiting during 24 hours) will be answered both at hospital admittance and discharge. For control patients the questionnaire will be answered at inclusion.
Other: 24 hours self-reported nutritional intake form — A nutritional intake form where relevant food and liquid items can be checked prospectively after consummation during 24 hours. This form will be filled in starting the morning following inclusion.

SUMMARY:
Nausea in early pregnancy (emesis gravidarum) is very common but most often self-limiting. Hyperemesis gravidarum; where nausea and vomiting is severe and protracted is potentially dangerous for the woman and her foetus and necessitates hospital treatment. An English questionnaire (PUQE; Pregnancy Unique Questionnaire of Emesis) exists that can differentiate between uncomplicated emesis and the severe hyperemesis condition. This questionnaire has been translated to Norwegian. The investigators want to test the ability of this questionnaire to differentiate the grade of nausea/vomiting between a group of presumed normal pregnant woman and patients treated for hyperemesis gravidarum in a Norwegian population. The investigators also want to relate the PUQE questionnaire scoring to the women/patients' self-reported nutritional intake during 24 hours.

DETAILED DESCRIPTION:
This is a prospective case-control study validating Pregnancy Unique Questionnaire of Emesis (PUQE) in a Norwegian population. The questionnaire has been translated from English to Norwegian by authorized translators. The Norwegian questionnaire's title is Svangerskaps Utløst Kvalme Kvantifisering (SUKK). The Norwegian version has been independently back-translated to English. The back-translated version has been approved by the original author Gideon Koren.

The primary objective is to evaluate if the questionnaire score is significantly different between a group of presumed healthy pregnant woman and a group of patients hospitalized with hyperemesis gravidarum.

The women will also fill in a self-reported 24-hours nutritional intake diary and this will be related to the Pregnancy Unique Questionnaire of Emesis (PUQE)score. For patients hospitalized with hyperemesis gravidarum the Pregnancy Unique Questionnaire of Emesis (PUQE)score both at admission and discharge will be compared.

Background clinical information for both groups at enrollment will be recorded as well as pregnancy outcome for woman and child.

The study has been approved by the Institutional Board as well as the Norwegian Regional Ethical Committee (REK Norway). Women will be included after giving informed written consent. Data will be stored electronically, anonymised, at a designated research server in accordance with the institutional research rules.

The sample size have been determined on basis of a similar study evaluating different nutritional status in emesis and hyperemesis patients, using 20 patients in each group. We aim to include 30 patients in each group.

Patients with diagnose of Hyperemesis gravidarum admitted form 1st of May 2013 will be consecutively asked to participate. Control patients will be recruited by invitation at primary care facilities or private out-patient gynaecologists.

Statistical analyses will be performed using Statistical Package for the Social Sciences (SPSS). Categorical variables will be compared using Chi-square test and continuous variables by non-parametric tests. Paired test will be used when comparing Pregnancy Unique Questionnaire of Emesis (PUQE)scores sequentially from admittance to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant healthy women (controls)
* Patients admitted to hospital for hyperemesis gravidarum

Exclusion Criteria:

* Pregnancy duration at inclusion more than 16 weeks
* Unable to understand and read/write Norwegian
* Conditions other than hyperemesis leading to nausea/vomiting

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Hyperemesis patients; recruited from university hospital clinic (normally 60 patients admitted during 12 months)
  Control paitients recruited from primary care/private practice out-patient gynaecologists
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy Unique Questionnaire of Emesis (PUQE) score reported by hyperemesis patients versus normal pregnant women | 24 hours after inclusion
  Pregnancy Unique Questionnaire of Emesis (PUQE) score range from 3 to 15. Scores reported for the first 24 hours after inclusion will be compared between hyperemesis patients and healthy pregnant control women

SECONDARY OUTCOMES:
Pregnancy Unique Questionnaire of Emesis (PUQE) score in relation to self reported 24 hours nutritional intake registration (estimated caloric intake)in hyperemesis patients versus normal pregnant women | 24 hours after inclusion
  The Pregnancy Unique Questionnaire of Emesis (PUQE) scores from hyperemesis and control women will be compared to self-reported 24 hours nutritional intake

OTHER OUTCOMES:
Change in Pregnancy Unique Questionnaire of Emesis (PUQE) score from hospital admittance to discharge | From hospital admission to discharge, mean 7 days
  Change in Pregnancy Unique Questionnaire of Emesis (PUQE) score for hyperemesis gravidarum patients from first assessment at hospital admission and again at hospital discharge
Pregnancy Unique Questionnaire of Emesis (PUQE) score at inclusion related to change in patient weight (kg)from start of pregnancy to inclusion for hyperemesis patients versus normal pregnant women | From pre-pregnancy to inclusion (mean 9 weeks pregnancy length)
  Change of weight (gain or loss) from pre-pregnant to time of inclusion related to Pregnancy Unique Questionnaire of Emesis (PUQE) scores for hyperemesis and control women
Change of Pregnancy Unique Questionnaire of Emesis (PUQE) score and patient weight (kg) | From inclusion to delivery (mean 7 months)
  Change of weight (gain or loss) from inclusion to time of delivery related to Pregnancy Unique Questionnaire of Emesis (PUQE) scores at inclusion for hyperemesis and control women
Pregnancy Unique Questionnaire of Emesis (PUQE) score related to the baby's weight (kg)in hyperemesis patients versus normal pregnant women | From inclusion to delivery (mean 7 months)
  Pregnancy Unique Questionnaire of Emesis (PUQE) scores at inclusion for hyperemesis versus control women is related to the baby's weight at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jone Trovik, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Dpt. of Obstetrics and Gynaecology, Haukeland University Hospital, Bergen, Hordaland
  - Dpt Obstetrics Gynaecology, Stavanger University Hospital, Stavanger, Rogaland

REFERENCES:
- [Background] Lacasse A, Rey E, Ferreira E, Morin C, Berard A. Validity of a modified Pregnancy-Unique Quantification of Emesis and Nausea (PUQE) scoring index to assess severity of nausea and vomiting of pregnancy. Am J Obstet Gynecol. 2008 Jan;198(1):71.e1-7. doi: 10.1016/j.ajog.2007.05.051. PMID 18166311
- [Background] Koren G, Piwko C, Ahn E, Boskovic R, Maltepe C, Einarson A, Navioz Y, Ungar WJ. Validation studies of the Pregnancy Unique-Quantification of Emesis (PUQE) scores. J Obstet Gynaecol. 2005 Apr;25(3):241-4. doi: 10.1080/01443610500060651. PMID 16147725
- [Background] van Stuijvenberg ME, Schabort I, Labadarios D, Nel JT. The nutritional status and treatment of patients with hyperemesis gravidarum. Am J Obstet Gynecol. 1995 May;172(5):1585-91. doi: 10.1016/0002-9378(95)90501-4. PMID 7755076